CLINICAL TRIAL: NCT03938935
Title: Repair of Flexor Tendon Injuries With Eight Strand Core Stitch Without Postoperative Splinting
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mina Micheal Anwer Fahmy (Other)
Responsible Party: Sponsor-Investigator, Mina Micheal Anwer Fahmy, Resident of Trauma and Orthopedic surgery-Assiut university, Assiut University
Organization: Assiut University (Other)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: Repair of flexor tendon injury
Record Dates: First submitted 2019-05-03; First posted 2019-05-06 (Actual); Last update posted 2019-05-07 (Actual); Status verified 2019-05

CONDITIONS: Flexor Tendon Repair

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Absorbable polydioxanone suture (PDS) — PDS is a Polydioxanone synthetic monofilament which is absorbable.

SUMMARY:
Evaluation of early active postoperative mobilisation in flexor tendon injuries without postoperative splinting

DETAILED DESCRIPTION:
Flexor tendon injuries are a common event as the tendons lie close to the skin and so are usually the result of either lacerations such as those from knives or glass, from crush injuries and occasionally they can rupture from where they are joined at the bone during contact sports such as football, rugby and wrestling. Flexor tendon injuries are a challenging problem for orthopaedic surgeons due to three main reasons. Firstly, flexor tendon injuries of the hands are a clinical problem because they cannot heal without surgical treatment, as the two ends need to be surgically brought together for the healing to occur unlike other tendons including the Achilles tendon where it could be placed into plantar flexion to heal. Secondly postoperative management needs to be carefully planned as mobilisation has shown to be essential to prevent adhesions and improve gliding but this can risk rupture. Lastly due to the unique anatomy of the tendons running through flexor tendon sheaths to function, surgeons need to plan preventing increasing the bulkiness of the tendon through its sheath, which is not always possible from scarring as this affects the functional outcome of the tendon

-_ The ultimate goal of surgical intervention has remained constant: to achieve enough strength to allow early motion, to prevent adhesions within the tendon sheath, and to restore the finger to normal range of motion and function.

* The successful repair requires minimal gapping at the repair site or interference with tendon vascularity, secure suture knots, smooth junction of tendon end and having sufficient strength for healing.
* The strength of the core suture is one of the important factors for valid flexor tendon repair. It is obvious that an increased strand number increases repair gap resistance and strength

ELIGIBILITY:
Inclusion Criteria:

1. Adult patient ( > 16 years)
2. Flexor tendon injuries zones (II,III,IV,V)

Exclusion Criteria:

1. Patients < 16 years
2. Flexor tendon injuries zone I

2- Fracture of hand,wrist or forearm bones 3- Associated nerve injuries

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Estimated)
Dates: Start 2019-10 (Estimated); Primary Completion 2021-02 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Early postoperative mobilisation of fingers (active & passive) - Follow up will be done according to DASH (Disability of arm,shoulder and hand) score at 6 weeks | one and half month

REFERENCES:
- [Background] Myer C, Fowler JR. Flexor Tendon Repair: Healing, Biomechanics, and Suture Configurations. Orthop Clin North Am. 2016 Jan;47(1):219-26. doi: 10.1016/j.ocl.2015.08.019. PMID 26614935